CLINICAL TRIAL: NCT04837053
Title: An Individualized Decision Aid for Physicians and Patients for Total Knee Replacement in Osteoarthritis (Value-based TKR): Study Protocol for a Multi-center, Stepped Wedge, Cluster Randomized Controlled Trial
Brief Title: Implementation of Indication Criteria for Total Knee Replacement in Osteoarthritis (Value-based TKR)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: Innovation Fund of the Joint Federal Committee (Gemeinsamer Bundesausschuss, G-BA), Germany (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Value-based TKR
Record Dates: First submitted 2021-02-22; First posted 2021-04-08 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Knee Osteoarthritis; Arthroplasty, Replacement, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Physicians

STUDY DESIGN:
Intervention Model Description: Pragmatic Multicenter Cluster Randomized Controlled Trial with stepped wedged design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention cluster (Experimental): EKIT tool
  Interventions: Other: Digital decision aid for physicians and patients
- Control Cluster (Active Comparator): routine care
  Interventions: Other: Routine care

INTERVENTIONS:
Other: Digital decision aid for physicians and patients — The intervention consists of three parts: (1) the EKIT tool provides a systematic presentation of individual patient and disease-specific information; (2) it visualizes the fulfilment of the indication criteria recommanded in corresponding german guideline; (3) it presents health information about total knee replacement.
  Arms: Intervention cluster
Other: Routine care — Care as usual within the included study sites.
  Arms: Control Cluster

SUMMARY:
The aim of this trial is to investigate the effect of a medical decision aid (EKIT-Tool) on decision quality for knee arthroplasty.

DETAILED DESCRIPTION:
The tool will guide the SDM process and support the consultation, providing a systematic presentation of individual patient and disease-specific information and the fulfilment of indication criteria. Furthermore, it will present health information about knee replacement to empower the patient. To investigate the effect of the tool on decision quality, we choose a prospective multi-center, stepped wedge, cluster randomized controlled trial (SW-RCT) design.

ELIGIBILITY:
Inclusion Criteria:

* patient with knee osteoarthritis who are candidates for knee replacement
* capacity to consent
* understanding of the German language (written and oral)
* age of 18 years or older
* informed consent

Exclusion criteria:

* meeting not all inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1092 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Decision quality | immediately after the intervention/procedure/surgery
  Decision quality measured by DQI-Knee Osteoarthritis v2.0

SECONDARY OUTCOMES:
Fulfillment of patient expectations | 12 months
  Fulfillment of patient expectations measured by a 5-point Likert-scale (not at all, no, unsure, yes partially, yes completely)
Oxford Knee Score (OKS) | 12 month
  Oxford Knee Score (0 worst to 48 best)

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Lützner, MD, Principal Investigator — TU Dresden
Locations (1):
- University Center of Orthopedics, Trauma and Plastic Surgery, University Hospital Carl Gustav Carus, Technische Universität Dresden, Dresden, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lange T, Deckert S, Beyer F, Hahn W, Einhart N, Roessler M, Sedlmayr M, Schmitt J, Lutzner J. An individualized decision aid for physicians and patients for total knee replacement in osteoarthritis (Value-based TKR study): study protocol for a multi-center, stepped wedge, cluster randomized controlled trial. BMC Musculoskelet Disord. 2021 Sep 12;22(1):783. doi: 10.1186/s12891-021-04546-5. PMID 34511058
- [Derived] Lutzner J, Deckert S, Beyer F, Hahn W, Malzahn J, Sedlmayr M, Gunther KP, Schmitt J, Lange T; Value-based Total Knee Replacement Study Group. Evaluation of a Digital Decision Aid for Knee Replacement Surgery. Dtsch Arztebl Int. 2024 Aug 23;121(17):566-572. doi: 10.3238/arztebl.m2024.0152. PMID 39109409